CLINICAL TRIAL: NCT00475566
Title: A Study to Evaluate the Safety and Performance of the Dynalink®-E, Everolimus Eluting Peripheral Stent System for Treating Atherosclerotic de Novo or Restenotic Native Superficial Femoral and Proximal Popliteal Artery Lesions
Brief Title: A Safety and Efficacy Study of the Dynalink®-E Everolimus Eluting Peripheral Stent System
Acronym: STRIDES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Marie-Helene Bettiol, Abbott Vascular
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06-103
Record Dates: First submitted 2007-05-16; First posted 2007-05-21 (Estimated); Last update posted 2011-03-10 (Estimated); Status verified 2011-03

CONDITIONS: Atherosclerosis; Peripheral Vascular Disease
MeSH Terms: conditions — Atherosclerosis; Peripheral Vascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Other): This is a prospective, non-randomized, single-arm, multi-center study. A projected 100 patients will receive the stent(s) in this study at approximately 10-15 European sites. The primary objective is to evaluate the safety and performance of the Dynalink®-E everolimus eluting peripheral stent system for the treatment of patients with atherosclerotic de novo or restenotic native superficial femoral or proximal popliteal lesions.
  Interventions: Device: Dynalink®-E everolimus-eluting peripheral stent; Device: Dynalink®-E, everolimus-eluting peripheral stent

INTERVENTIONS:
Device: Dynalink®-E everolimus-eluting peripheral stent — Stenting of atherosclerotic de novo or restenotic lesions (> 50% stenosis) in the native superficial femoral or proximal popliteal artery
Device: Dynalink®-E, everolimus-eluting peripheral stent — Stenting of atherosclerotic de novo or restenotic lesions (> 50% stenosis) in the native superficial femoral or proximal popliteal artery

SUMMARY:
The purpose of this first-in-man study is to evaluate the safety and performance of the Dynalink®-E everolimus eluting peripheral stent system for the treatment of patients with atherosclerotic de novo or restenotic native superficial femoral and proximal popliteal lesions.

Abbott Vascular is ceasing data analysis of the STRIDES Clinical Trial after 2 years. The decision to discontinue the study is not related to any safety concern. The rationale for this proposal is based on the following considerations:

The performance of DYNALINK-E from STRIDES shows no device- or procedure-related deaths and no stent fractures, and the rate of additional revascularizations has been stable since approximately 14 months after the procedure.

Evaluations of the bare metal nitinol DYNALINK and ABSOLUTE stents in the clinical literature show low rates of death, reintervention and stent fracture, which are consistent with STRIDES and demonstrate the safety of the nitinol stent platform of the DYNALINK-E.

Long-term animal studies show no concerns with the drug or polymer coating of DYNALINK-E - everolimus tissue concentration drops below the quantifiable limit by approximately 17 months after implant, and vascular response to the coating is normal with widely patent lumens and struts incorporated into vessel tissue.

The safety and performance of the DYNALINK-E has been substantiated by its clinical and pre-clinical data, and by the clinical data of similar products. Given the demonstrated mechanical integrity of the stent along with the evidence of a healthy long-term vascular response, there is a reasonable expectation of continued low event rates.

DETAILED DESCRIPTION:
A prospective, Non-Randomized, Single-arm, Multi-center, Clinical Study to Evaluate the Safety and Performance of the Dynalink®-E, Everolimus Eluting Peripheral Stent System for the Treatment of Atherosclerotic de Novo or Restenotic Native Superficial Femoral and Proximal Popliteal Artery Lesions.

ELIGIBILITY:
Inclusion Criteria:

* Rutherford Becker Category 2-5
* Single de novo or restenotic lesion in the superficial femoral or proximal popliteal artery
* Disease segment length 30-170 mm
* >50% diameter stenosis or total occlusion
* Target reference vessel diameter 4.3-7.3 mm

Exclusion Criteria:

* Target lesion previously treated with stent or surgery
* Rutherford Becker Category 0, 1, or 6
* Immunosuppressive disorder or currently receiving immunosuppressive agents
* Serum creatinine >2.5 mg/dl

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2007-05; Primary Completion 2008-07 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
In-stent binary restenosis (>50% stenosis), as measured by duplex ultrasound | 6 months

SECONDARY OUTCOMES:
Angiographic in-stent binary restenosis rate (>50%) | 12 months
Angiographic mean in-stent late loss, in-stent mean minimum lumen diameter (MLD), percent diameter stenosis | 12 months
Primary, and secondary patency | 1, 6, 12, 18 months, 2, 3, 4, 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Johannes Lammer, M.D., Principal Investigator — Allgemeines Krankenhaus der Stadt Wien
Locations (10):
- Austria (2):
  - Landeskrankenhaus Klagenfurt, Klagenfurt
  - Allgemeines Krankenhaus der Stadt Wien- AKH Wien, Vienna
- Belgium (3):
  - Sint Blasius Hospital, Dendermonde
  - ZOL St. Jan, Ghent
  - University Hospital, Ghent
- Germany (4):
  - Herzzentrum Bad Krozingen, Bad Krozingen
  - The Jewish Hospital Berlin, Berlin
  - Herzzentrum Leipzig, Leipzig
  - University Hospital Tübingen, Tübingen
- Casa di Cura di Montevergine, Mercogliano, Italy

REFERENCES:
- [Derived] Lammer J, Scheinert D, Vermassen F, Koppensteiner R, Hausegger KA, Schroe H, Menon RM, Schwartz LB. Pharmacokinetic analysis after implantation of everolimus-eluting self-expanding stents in the peripheral vasculature. J Vasc Surg. 2012 Feb;55(2):400-5. doi: 10.1016/j.jvs.2011.08.048. Epub 2011 Nov 1. PMID 22051872
- [Derived] Lammer J, Bosiers M, Zeller T, Schillinger M, Boone E, Zaugg MJ, Verta P, Peng L, Gao X, Schwartz LB. First clinical trial of nitinol self-expanding everolimus-eluting stent implantation for peripheral arterial occlusive disease. J Vasc Surg. 2011 Aug;54(2):394-401. doi: 10.1016/j.jvs.2011.01.047. Epub 2011 Jun 12. PMID 21658885